CLINICAL TRIAL: NCT01500889
Title: Comparative Study of Conventional Lateral Internal Sphincterotomy, V-Y Anoplasty and Tailored Lateral Internal Sphincterotomy With V-Y Anoplasty in Treatment of Chronic Anal Fissure
Brief Title: Conventional Lateral Internal Sphincterotomy, V-Y Anoplasty and Tailored Lateral Internal Sphincterotomy With V-YF in Treatment of Chronic Anal Fissure(CAF)
Acronym: CAF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Alaa Magdy, Faculity of medicine, mansoura university, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: anal fissure
Record Dates: First submitted 2011-12-15; First posted 2011-12-29 (Estimated); Last update posted 2011-12-29 (Estimated); Status verified 2011-12

CONDITIONS: Chronic Anal Fissure
Keywords: Anal fissure; Advancement flap; Internal sphincterotomy
MeSH Terms: conditions — Fissure in Ano | interventions — gene 11 protein, Rotavirus B

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CLI sphincterotomy (Active Comparator): Conventional Lateral internal sphincterotomy LIS was performed in the lithotomy position by a standard open technique, briefly; a 5-mm incision was made into the perianal skin along the intersphinteric groove. The internal anal sphincter was then dissected and a segment withdrawn with a pair of artery forces and divided with diathermy to the level of the dentate line. Figures 5, 6, 7 and 8 illustrate the procedure.
  Interventions: Procedure: Group I: Conventional Lateral internal sphincterotomy:
- GroupII: V-Y advancement flap (Active Comparator): The V-Y advancement flap was performed by making a V-shaped incision from the edges of the fissure extending about 4 cm from the anal verge and away from the midline. The V-shaped flap formed of skin and subcutaneous fat was mobilized sufficiently to allow advancement into the anal canal to cover the fissure defect. Care was taken to preserve enough pedicles to ensure adequate blood supply. The base of flap was sutured to the lower anal mucosa with interrupted 000 Vicryl Rapide. Figures 1, 2, 3 and 4 illustrate the procedure.
  Interventions: Procedure: GroupII: V-Y advancement flap
- TLIS with VY anoplasty (Active Comparator): Tailored lateral sphincterotomy was performed in the lithotomy position by a standard open technique, briefly; a 5-mm incision was made into the perianal skin along the intersphinteric groove. The internal anal sphincter was then dissected and a segment withdrawn with a pair of artery forces and divided with diathermy, the extent of sphincterotomy was done to be more or less equal to the length of the fissure. Then the V-Y advancement flap was performed.
  Interventions: Procedure: GroupIII: Tailored LIS with V-Y advancement flap

INTERVENTIONS:
Procedure: Group I: Conventional Lateral internal sphincterotomy: — LIS was performed in the lithotomy position by a standard open technique, briefly; a 5-mm incision was made into the perianal skin along the intersphinteric groove. The internal anal sphincter was then dissected and a segment withdrawn with a pair of artery forces and divided with diathermy to the level of the dentate line. Figures 5, 6, 7 and 8 illustrate the procedure.
  Other Names: Group 1
  Arms: CLI sphincterotomy
Procedure: GroupII: V-Y advancement flap — GroupII: V-Y advancement flap:
  The V-Y advancement flap was performed by making a V-shaped incision from the edges of the fissure extending about 4 cm from the anal verge and away from the midline. The V-shaped flap formed of skin and subcutaneous fat was mobilized sufficiently to allow advancement into the anal canal to cover the fissure defect. Care was taken to preserve enough pedicles to ensure adequate blood supply. The base of flap was sutured to the lower anal mucosa with interrupted 000 Vicryl Rapide.
  Other Names: Group 11
  Arms: GroupII: V-Y advancement flap
Procedure: GroupIII: Tailored LIS with V-Y advancement flap — Tailored lateral sphincterotomy was performed in the lithotomy position by a standard open technique, briefly; a 5-mm incision was made into the perianal skin along the intersphinteric groove. The internal anal sphincter was then dissected and a segment withdrawn with a pair of artery forces and divided with diathermy, the extent of sphincterotomy was done to be more or less equal to the length of the fissure. Then the V-Y advancement flap was performed.
  Other Names: Group III
  Arms: TLIS with VY anoplasty

SUMMARY:
The investigators compared conventional lateral internal sphincterotomy (CLIS), V-Y anal flap, and combined tailored lateral internal sphincterotomy with V-Y anal flap (TLIS with V-YF) in a randomized prospective study in patients undergoing treatment for chronic anal fissure.

DETAILED DESCRIPTION:
Group I: Conventional Lateral internal sphincterotomy:

LIS was performed in the lithotomy position by a standard open technique, briefly; a 5-mm incision was made into the perianal skin along the intersphinteric groove. The internal anal sphincter was then dissected and a segment withdrawn with a pair of artery forces and divided with diathermy to the level of the dentate line. Figures 5, 6, 7 and 8 illustrate the procedure.

GroupII: V-Y advancement flap:

The V-Y advancement flap was performed by making a V-shaped incision from the edges of the fissure extending about 4 cm from the anal verge and away from the midline. The V-shaped flap formed of skin and subcutaneous fat was mobilized sufficiently to allow advancement into the anal canal to cover the fissure defect. Care was taken to preserve enough pedicles to ensure adequate blood supply. The base of flap was sutured to the lower anal mucosa with interrupted 000 Vicryl Rapide. Figures 1, 2, 3 and 4 illustrate the procedure.

GroupIII: Tailored lateral internal sphincterotomy with V-Y advancement flap:

Tailored lateral sphincterotomy was performed in the lithotomy position by a standard open technique, briefly; a 5-mm incision was made into the perianal skin along the intersphinteric groove. The internal anal sphincter was then dissected and a segment withdrawn with a pair of artery forces and divided with diathermy, the extent of sphincterotomy was done to be more or less equal to the length of the fissure. Then the V-Y advancement flap was performed All assessments were conducted by investigators who were blinded to the experimental condition. The primary outcome was complete healing (complete epithelization scare or no sign of fissure, healing was considered to be delayed if the wound had not completely healed by 6 weeks after the procedure). Secondary outcomes were operative time, length of hospital stay, anal incontinence (determined by Pescatori scoring system (32), time of relieve of pain, postoperative anal manometery, complications (eccyhmosis, haematoma, infection, disruption of flap, flap necrosis), persistent symptoms, patients satisfaction ( assessed on a visual analogue scale VAS), recurrence rate and quality of life.

Quality of life was assessed using the Gastrointestinal Quality of Life Index (GIQLI) developed by Eypasch and coworkers

ELIGIBILITY:
Inclusion Criteria:

* consecutive patients who treated for chronic anal fissure at colorectal surgery unite of Mansoura university hospital, Mansoura, Egypt.
* all patients were selected to have increased resting anal pressure above the upper limit of normal range.

Exclusion Criteria:

* patients with acute fissure
* patients who had resting anal pressure within the normal range or less than the normal
* cicatricial deformation
* large sentinel pile
* inflammatory bowel disease hemorrhoids
* fistula in ano and anal abscesses
* those who had undergone previous surgical procedure in the anal canal
* age above 80 years
* vascular disease
* scleroderma
* malnutrition
* coagulopathy

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2009-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
complete healing (complete epithelization scare or no sign of fissure, healing was considered to be delayed if the wound had not completely healed by 6 weeks after the procedure). | 1 year
  complete healing (complete epithelization scare or no sign of fissure, healing was considered to be delayed if the wound had not completely healed by 6 weeks after the procedure).

SECONDARY OUTCOMES:
Secondary outcomes were operative time | 1 year
  Secondary outcomes were operative time, length of hospital stay, anal incontinence (determined by Pescatori scoring system (32), time of relieve of pain, postoperative anal manometery, complications (eccyhmosis, haematoma, infection, disruption of flap, flap necrosis), persistent symptoms, patients satisfaction ( assessed on a visual analogue scale VAS), recurrence rate and quality of life.
length of hospital stay | one month
  early postoperative hospital stay
anal incontenance | one year
  using pescatori scoring
recurrence rate | one year
  recurrence rate
postoperative anal manometery | one year
  resting anal pressure
complication | one month
  necrosis, infection

CONTACTS AND LOCATIONS:
Overall Officials: Alae magdy, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Result] Littlejohn DR, Newstead GL. Tailored lateral sphincterotomy for anal fissure. Dis Colon Rectum. 1997 Dec;40(12):1439-42. doi: 10.1007/BF02070709. PMID 9407982
- [Result] Chambers W, Sajal R, Dixon A. V-Y advancement flap as first-line treatment for all chronic anal fissures. Int J Colorectal Dis. 2010 May;25(5):645-8. doi: 10.1007/s00384-010-0881-1. Epub 2010 Feb 23. PMID 20177691
- [Result] Giordano P, Gravante G, Grondona P, Ruggiero B, Porrett T, Lunniss PJ. Simple cutaneous advancement flap anoplasty for resistant chronic anal fissure: a prospective study. World J Surg. 2009 May;33(5):1058-63. doi: 10.1007/s00268-009-9937-1. PMID 19225835
- [Result] Hancke E, Rikas E, Suchan K, Volke K. Dermal flap coverage for chronic anal fissure: lower incidence of anal incontinence compared to lateral internal sphincterotomy after long-term follow-up. Dis Colon Rectum. 2010 Nov;53(11):1563-8. doi: 10.1007/DCR.0b013e3181f0869f. PMID 20940607
- See also: Mansoura University — http://www.mans.edu.eg